CLINICAL TRIAL: NCT05042687
Title: Comparative Performance of Molecular Breast Imaging (MBI) to Magnetic Resonance Imaging (MRI) of the Breast in Identifying and Excluding Breast Carcinoma in Women at High Risk for Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-0927; NCI-2021-09605 (Other: NCI CTRP Clinical Trials Registry)
Record Dates: First submitted 2021-08-25; First posted 2021-09-13 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Technetium Tc 99m Sestamibi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tc99m sestamibi (Experimental): MBI uses an injection of a small amount of radioactive material called technetium99m (Tc99m) sestamibi
  Interventions: Drug: Tc99m sestamibi

INTERVENTIONS:
Drug: Tc99m sestamibi — Given by IV

SUMMARY:
To evaluate the diagnostic performance of Tc99m sestamibi (MBI) compared to breast MRI in women who are at high risk for developing breast cancer.

To assess the relationship of tumor size, histologic subtype and location of lesion and how it affects lesion conspicuity and sensitivity in MBI detected cancers.

DETAILED DESCRIPTION:
Primary Objective:

-To compare the diagnostic performance of Molecular Breast Imaging (MBI) to breast Magnetic Resonance Imaging (MRI) in women who are at high risk of developing breast cancer.

Secondary Objectives:

* To evaluate the sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of MBI compared to breast MRI in women who are at high risk of developing breast cancer.
* To assess patient preference for the two examinations by conducting a post examination survey and follow up questionnaire (see addendum).
* To assess the relationship of tumor size, histologic subtype and location of lesion with lesion conspicuity (mild, moderate, marked uptake compared to background activity) according to MBI lexicon [1].

ELIGIBILITY:
Inclusion Criteria:

* The subjects to be studied will include female patients ages 18 and older of any race, identified as carrying an elevated risk for breast cancer referred to MDACC.
* High risk may be defined as having a calculated lifetime risk >20%, histopathology of lobular neoplasia or atypical ductal hyperplasia, atypia NOS or a genetic mutation known to predispose the patient to breast cancer.
* Subject who are scheduled for a Breast MRI who are willing to participate fully in all aspects of the study including completing both a Breast MRI & MBI screening exam within a two-week time window, a biopsy of any positive findings and complete a post examination survey. Consent for the enrollment may be obtained upon scheduling the MRI examination. For non-English speakers, a language interpreter will assist in translation.
* Written consent will be obtained from all participants to obtain MBI of the breasts and biopsy as indicated, based on findings. All participants will be asked to provide a post examination survey of their experience with both tests.

Exclusion Criteria:

* Subjects who are pregnant will be excluded as MBI exam involves injection of radioactive tracer
* contrast enhanced MRI involves gadolinium injection, both of which are contraindicated during pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 300 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To establish the diagnostic performance of Molecular Breast Imaging (MBI) to breast Magnetic Resonance Imaging (MRI) in women who are at high risk of developing breast cancer | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Adrada, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org